CLINICAL TRIAL: NCT02756455
Title: Procalcitonin Reveals Early Dehiscence In Gastric Surgery: the PREDIGS Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Valentina Giaccaglia, MD, University of Roma La Sapienza
Other Study IDs: PREDIGS
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; procalcitonin
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- gastric cancer pts undergoing surgery: all pts receiving gastric resection for cancer, with anastomosis
  Interventions: Other: gastric cancer pts undergoing surgery

INTERVENTIONS:
Other: gastric cancer pts undergoing surgery — Measure PCT (procalcitonin), CRP (C-reactive protein) and WBC (white blood cell count) in 3rd and 5th postoperative day and registration of all intra and postoperative complications

SUMMARY:
Background. Gastric cancer surgery is associated with high risk for postoperative morbidity and mortality. Anastomotic leak (AL) is one of the worst complications associated with relevant short and long-term sequelae. Procalcitonin (PCT) is a biomarker used to monitor bacterial infections and guide antibiotic therapy and has been shown to have better predictive value of AL after colorectal surgery than C-reactive protein (CRP) and white blood cell count (WBC).

Purpose. Investigators designed a monocentric pilot study to test if PCT might be a sensitive and reliable marker of AL after gastric surgery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing all different kinds of gastric surgery (from partial to total gastrectomy) for cancer, WITH an anastomosis performed
* elective setting

Exclusion Criteria:

* age < 18 years
* pregnant women
* patients undergoing gastric surgery for benign disease or other kinds of gastric surgery without an anastomosis being performed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing gastric cancer surgery in our institution
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
% of patients with leaks after gastric surgery correctly identified by the biomarkers (PCT and CRP) | 2 years
  PCT: procalcitonin, CRP: C-reactive protein
% of patients without leaks after gastric surgery correctly identified by PCT and CRP | 2 years
  PCT: procalcitonin, CRP: C-reactive protein

SECONDARY OUTCOMES:
PCT cut-off that gives good negative predictive (NPV) value for leak after gastric surgery in 3rd POD | 2 years
  procalcitonin (PCT) cuts-off in 3rd post-operative day (POD) with a good NPV
PCT cut-off that gives good negative predictive value for leak after gastric surgery in 5th POD | 2 years
  PCT cuts-off in 5th POD with a good NPV

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Andrea University Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No